CLINICAL TRIAL: NCT05269771
Title: Treatment Plan for Managed Access Program (MAP) to Provide Access to Ruxolitinib, for Patients With Polycythemia Vera (PV)
Brief Title: MAP to Provide Access to Ruxolitinib, for Patients With Polycythemia Vera
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CINC424B2002I
Record Dates: First submitted 2022-02-16; First posted 2022-03-08 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Polycythemia Vera
Keywords: INC424; Ruxolitinib; Jakavi; MAP; Manage access program
MeSH Terms: conditions — Polycythemia Vera | interventions — ruxolitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Ruxolitinib — Patients may self-administer daily ruxolitinib tablets qd or bid orally, without regard to food, in accordance with specified dosing schedule provided by the investigator.
  Other Names: Jakavi

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to ruxolitinib for eligible patients diagnosed with Polycythemia Vera. The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

DETAILED DESCRIPTION:
The requesting Treating Physician must submit a request for access to drug (often referred to as Compassionate Use) to Novartis which will review and approve by the medical team experienced with the drug and indication.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this Treatment Plan have to meet all of the following criteria:

1. Male or female aged 12 or over
2. Confirmed diagnosis of PV based on World Health Organization (WHO) criteria
3. Patients must have a treatment history for PV that meets the definition of resistance or intolerance to hydroxyurea (HU) or other cytoreductive therapy
4. Patients with a peripheral blood blast count of 0% at screening
5. Patients must have recovered or stabilized sufficiently from adverse drug reactions associated with prior treatments before beginning treatment with ruxolitinib
6. Patients with an Eastern Cooperative Oncology Group (ECOG) score of 0, 1 or 2 Written patient informed consent must be obtained prior to start of treatment.

Exclusion Criteria:

Patients eligible for this Treatment Plan must not meet any of the following criteria:

1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as ruxolitinib.
2. Presence of an active uncontrolled infection including significant bacterial, fungal, viral (including CMV, EBV, HHV-6, HBV, HCV, BK or HIV) or parasitic infection requiring treatment. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection. Patients with inactive chronic infection (without viral replication) can be enrolled.
3. History of progressive multifocal leuko-encephalopathy (PML).
4. Presence of severely impaired renal function defined by serum creatinine > 2 mg/dL (>176.8 μmol/L), or have estimated creatinine clearance < 30 ml/min measured or calculated by Cockroft Gault equation.
5. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, UNLESS they are

   * women whose sexual orientation precludes intercourse with a male partner.
   * women whose partners have been sterilized by vasectomy or other means.
   * using a highly effective method of birth control (i.e. one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices (IUDs); periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable throughout the period of treatment and 30 days after treatment discontinuation.

   Any female aged 8 years and above is to be treated as a woman of child-bearing potential.

   Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
6. Pregnancy
7. Not able to understand and to comply with treatment instructions and requirements

Ages: 12 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- Novartis Investigative Site, Orange, New South Wales, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Calgary, Alberta, Canada
- Novartis Investigative Site, Tehran, Iran
- Israel (5):
  - Novartis Investigative Site, Kfar Saba, Israel
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Rehovot
  - Novartis Investigative Site, Tel Aviv
  - Novartis Investigative Site, Tel Giborim Holon
- Novartis Investigative Site, Groningen, Netherlands
- Poland (6):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wałbrzych
  - Novartis Investigative Site, Wroclaw
- United Kingdom (6):
  - Novartis Investigative Site, Hereford
  - Novartis Investigative Site, Kent
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Poole
  - Novartis Investigative Site, Salisbury